CLINICAL TRIAL: NCT02973568
Title: Comparative Study on Acute Pain Evaluation Between Spanish and French Hospital Emergency Unit
Acronym: DASAU
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Collaborators: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Other Study IDs: DASAU
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2016-11

CONDITIONS: Pain; EMERGENCY MEDICINE
MeSH Terms: conditions — Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational Study

SUMMARY:
Today, pain is a difficult affordable subject in Spain. There are however 187 units of pain care with a consultations rate in emergency center of more than 60%.For example OXYCODONE(opioid analgesic)is widely used while it's under used in Spain.

In the same way MEOPA(Kalinox) is a new approach of pain care daily used as well in France (for example in dislocated shoulder pain, or ulceration care...etc) There are lots of studies relative to chronic pain but not too much about acute pain in Spain.That's why we want to focus our study on evaluation of acute pain treatment and efficacy in french and spanish hospital

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in emergency center for acute pain.
* Patient who accept to participate.

Exclusion Criteria:

* Refusal of patient to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Evety patient admitted in emergency center during 1 month for acute pain and who need treatment for pain
Sampling Method: Non-Probability Sample
Enrollment: 641 (Actual)
Dates: Start 2016-04-01; Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
pain VAS (visual analogic scale) | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Jonay PERERA GIL, PhD student, Study Director — Groupe Hospitalier Paris Saint-Joseph (FRANCE); Olivier GANANSIA, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided